CLINICAL TRIAL: NCT06653725
Title: Exogenous KETOne Supplements in Patients Hospitalized for Acute Heart Failure. A Randomized Clinical Trial (KETO-AHF)
Brief Title: Exogenous KETOne Supplements in Patients Hospitalized for Acute Heart Failure
Acronym: KETO-AHF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Viborg Regional Hospital (Other); Hospitalsenhed Vest, Herning (Unknown); Odense University Hospital (Other); Aalborg University Hospital (Other); Rigshospitalet, Denmark (Other); Copenhagen University Hospital at Herlev (Other); Amager Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KETO-AHF; 1-10-72-63-24 (Registry Identifier: De videnskabsetiske Komitéer for Region Midtjylland)
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-09

CONDITIONS: Acute Heart Failure (AHF)
Keywords: Acute heart failure; Ketone supplements; Ketones; 3-hydroxybutyrate; 1,3-butanediol; six-minute walk test; win ratio
MeSH Terms: conditions — Ketosis | interventions — 1,3-butylene glycol

STUDY DESIGN:
Intervention Model Description: Patients are randomized 1:1 to 1,3-butanediol or matching placebo treatment for 30 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1,3-butanediol (Experimental): 1,3-butanediol (Ketone-IQ®) 118 mL (33 g) servings trice daily
  Interventions: Dietary Supplement: 1,3-butanediol
- Placebo (Placebo Comparator): Taste-matched placebo (isovolumic, isoviscous water with stevia) 118 mL servings trice daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 1,3-butanediol — 1,3-butanediol (Ketone-IQ®) 118 mL (33 g) servings trice daily
  Arms: 1,3-butanediol
Dietary Supplement: Placebo — Taste-matched placebo (isovolumic, isoviscous water with stevia) 118 mL servings trice daily
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled trial to investigate the clinical efficacy of treatment with exogenous dietary ketone supplement containing 1,3-butanediol in patients hospitalized with acute heart failure (AHF), potentially leading to better clinical outcomes.

DETAILED DESCRIPTION:
Acute heart failure (AHF) is life-threatening with a 30-day mortality rate between 10% and 50%, especially in patients with cardiogenic shock. Current medical treatments have not shown a survival benefit in randomized trials, highlighting the need for new therapies. Ketone bodies, particularly 3-hydroxybutyrate (3-OHB), are vital for energy in the heart and brain during stress. Elevated 3-OHB levels from exogenous sources, such as ketone esters or 1,3-butanediol, enhance organ perfusion and improve cardiac function. In chronic heart failure (HF), 3-OHB infusion increases cardiac output and left ventricular ejection fraction (LVEF) without excess oxygen consumption, supporting its role as an efficient energy source. Short-term ketone ester treatment has been shown to improve hemodynamics, reduce NT-proBNP, and enhance physical performance in heart failure with reduced ejection fraction (HFrEF) patients. In AHF patients, ketone ester improved cardiac output, LVEF, and filling pressures. Emerging evidence suggests that 1,3-butanediol supplements may sustain ketosis longer, offering potential for practical dosing in the acute phase of heart failure.

This proposal aims to study the clinical efficacy of treatment with exogenous dietary ketone supplement containing 1,3-butanediol in patients hospitalized with AHF.

The primary hypothesis is that in patients hospitalized with AHF, a 30-day treatment with 1,3- butanediol has beneficial clinical effects as compared with placebo. Clinical benefit is defined as a hierarchical composite of death, heart failure (HF) events, change from baseline in the 6-minute walk test (6MWT), and change from baseline in NT-proBNP at 30 days, as assessed using win ratio statistics.

ELIGIBILITY:
The study will enroll adult patients (≥18 years) admitted with AHF as the primary diagnosis, meeting all the following criteria:

1. Documented new or worsening symptoms due to heart failure with at least one of the following: persistent dyspnea at rest or with minimal exertion, or fatigue.
2. Objective evidence of worsening heart failure, consisting of at least two physical examination findings consistent with fluid retention and/or end-organ hypoperfusion or one physical examination finding and at least one laboratory criterion:

   a) Physical examination findings considered to be due to heart failure, including new or worsened: i. Peripheral edema ii. Increasing abdominal distention or ascites (in the absence of primary hepatic disease) iii. Pulmonary rales/crackles/crepitations iv. Increased jugular venous pressure and/or hepatojugular reflux v. S3 gallop vi. Clinically significant or rapid weight gain thought to be related to fluid retention b) Laboratory evidence of worsening HF, if obtained within 24 hours of presentation, including: i. Increased B-type natriuretic peptide (BNP) / N-terminal pro-BNP (NT-proBNP) concentrations consistent with decompensation of heart failure. In patients with chronically elevated natriuretic peptides, an increase of >30% above baseline should be noted.

   ii. Radiological evidence of pulmonary congestion iii. Echocardiographic criteria include: Dilated inferior vena cava with minimal collapse on inspiration; decreased left ventricular outflow tract (LVOT) minute stroke distance (velocity time integral [VTI]); septal or lateral E/e' >15 or >12, respectively; D-dominant pulmonary venous inflow pattern.

   iv. Invasive diagnostic evidence with right heart catheterization showing a pulmonary capillary wedge pressure ≥18 mmHg, central venous pressure ≥12 mmHg, or a cardiac index <2.2 L/min/m2
3. Treatment with at least 40 mg of intravenous furosemide or its equivalent and/or intravenous vasoactive drugs and/or inotropic drugs.
4. An LVEF of ≤35% is required, measured during the present hospitalization.
5. Participants must present with elevated levels of natriuretic peptides, specifically NT-proBNP ≥600 pg/mL or BNP ≥150 pg/mL. For those in atrial fibrillation at the time of inclusion, NT-proBNP levels must be ≥900 pg/mL or BNP ≥225 pg/mL.

The enrollment window extends to the first five days of the hospital stay.

Exclusion Criteria:

1. Current hospitalization for AHF triggered by significant arrhythmia (atrial fibrillation/flutter with sustained ventricular response >110 beats per minute, clinically significant bradycardia, or sustained ventricular tachycardia)
2. Cardiogenic shock in INTERMACS level 1 or 2 (i.e. unstable hemodynamics despite inotropic/vasopressor therapy)
3. Likelihood or current use of mechanical circulatory support
4. Recent cardiac surgery within 3 days
5. Ongoing severe infection or sepsis, severe anemia, acute exacerbation of chronic obstructive pulmonary disease, pulmonary embolism, or cerebrovascular accident
6. Significant primary valvular disease (hemodynamically severe uncorrected primary cardiac valvular disease)
7. Planned implantation of a cardiac resynchronization therapy device
8. eGFR <15 mL/min/1.73 m2 during current hospitalization (unless ongoing continuous renal replacement therapy) or recurring dialysis
9. Known obstructive hypertrophic cardiomyopathy, congenital heart disease, acute mechanical cause of acute heart failure (e.g., papillary muscular rupture), acute myocarditis, or constrictive pericarditis according to the treating physician
10. Type 1 diabetes
11. Advanced liver disease (Child-Pugh class C)
12. Dementia or other cognitive disorder making the patient unable to give informed consent
13. Pregnancy or breastfeeding
14. Inability to intake oral substances or severe dysphagia
15. Significant gastrointestinal disease (i.e. severe inflammatory bowel disease or gastric ulcer)
16. Adherent to a ketogenic diet within 30 days of enrollment
17. Awaiting cardiac transplantation
18. Very severe lung disease and/or treatment with continuous home oxygen therapy
19. Major comorbidity, medical condition, or health issue that, according to the investigator's judgment, would hinder the participant's capacity to engage in or successfully finish the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in clinical benefit during 1,3-butanediol treatment versus placebo | From baseline (day 0) to end of treatment (day 30)
  Clinical benefit is defined through a hierarchical composite endpoint, using a win ratio, from day 0 to 30 in all-cause death and time to death, number of and time to heart failure events, ≥30 meters increase in the change from baseline to follow-up at 30 days in the 6MWT, (iv) >30% decrease in the change from baseline to follow-up at 30 days in NT-proBNP, and (v) % decrease in NT-proBNP (continuous variable).
  The primary endpoint will be evaluated using a win ratio, in an intention-to-treat approach, with participants analyzed within the treatment groups to which they were originally randomized. The win ratio method involves a pairwise hierarchical comparison of each participant against all others and is determined by dividing the total number of wins achieved by participants in the 1,3-butanediol group by the total number of losses.

SECONDARY OUTCOMES:
Time to all-cause death | From baseline (day 0) to end of treatment (day 30)
Time to first heart failure event | From baseline (day 0) to end of treatment (day 30)
Change in six-minute walking distance | From baseline (day 0) to end of treatment (day 30)
Change in daily activity level | From discharge, day 30, and end of treatment (day 30)
  When discharged, a wearable triaxial accelerometer will be placed around the wrist of the patient. The accelerometer will measure daily physical activity (milligravitational units) between discharge and 30-day follow-up.
Change in NT-proBNP | From baseline (day 0) to discharge and end of treatment (day 30)
Change in KCCQ-12 total summary score | From baseline (day 0) to discharge and end of treatment (day 30)
Change in VAS dyspnea score | From baseline (day 0) to discharge and end of treatment (day 30)
Change in physical exertion score during six- minute walk test | From baseline (day 0) to discharge and end of treatment (day 30)
Change in systolic blood pressure | From baseline (day 0) to discharge and end of treatment (day 30)
Change in body weight | From baseline (day 0) to discharge and end of treatment (day 30)
Diuretic response | From baseline (day 0) to discharge and end of treatment (day 30)
  Diuretic response will be defined as Δ weight kg/[(total intravenous dose)/40mg] + [(total oral dose)/80mg)] furosemide or equivalent loop diuretic dose
Cumulative dose of loop diuretic medication | From baseline (day 0) to discharge and end of treatment (day 30)
Need for inotropes | From baseline (day 0) to end of treatment (day 30)
Transfer to the intensive care unit | From baseline (day 0) to end of treatment (day 30)
Need for dialysis | From baseline (day 0) to end of treatment (day 30)

OTHER OUTCOMES:
Length of index hospital stay | From baseline (day 0) to end of treatment (day 30)
Days alive out of hospital | From baseline (day 0) to end of treatment (day 30)
Subject experiencing improvement/deterioration in NYHA Class | From baseline (day 0) to discharge, day 30, and end of treatment (day 30)
Change in estimated glomerular filtration rate | From baseline (day 0) to discharge and end of treatment (day 30)
  Pre-Specified Renal sub study
Change in hematocrit | From baseline (day 0) to discharge and end of treatment (day 30)
  Pre-Specified Renal sub study
Change in urine sodium | From baseline (day 0) to discharge and end of treatment (day 30)
  Pre-Specified Renal sub study
Change in urine 3-OHB | From baseline (day 0) to discharge and end of treatment (day 30)
  Pre-Specified Renal sub study
Change in insulin sensitivity | From baseline (day 0) to discharge and end of treatment (day 30)
  Pre-Specified Metabolic sub study
Change in cholesterol level | From baseline (day 0) and end of treatment (day 30)
  Pre-Specified Metabolic sub study
Change in left atrial volume | From baseline (day 0) and end of treatment (day 30)
  Pre-Specified Hemodynamic sub study
Change in LV filling pressure (E/e ́) | From baseline (day 0) and end of treatment (day 30)
  Pre-Specified Hemodynamic sub study
Change in LVEF | From baseline (day 0) and end of treatment (day 30)
  Pre-Specified Hemodynamic sub study
Change in LV end-systolic volume | From baseline (day 0) and end of treatment (day 30)
  Pre-Specified Hemodynamic sub study
Change in LV end-diastolic volume | From baseline (day 0) and end of treatment (day 30)
  Pre-Specified Hemodynamic sub study

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer Berg-Hansen, MD, PhD, Principal Investigator — Department of Cardiology, Aarhus University Hospital
Locations (8):
- Denmark (8):
  - Department of Cardiology, Aalborg University Hospital, Aalborg
  - Department of Cardiology, Aarhus University Hospital, Aarhus N
  - Department of Cardiology, Herlev-Gentofte Hospital, Copenhagen
  - Department of Cardiology, Rigshospitalet, Copenhagen
  - Department of Cardiology, Gødstrup Hospital, Herning, Denmark, Herning
  - Department of Cardiology, Copenhagen University Hospital - Amager and Hvidovre Hospital, Hvidovre
  - Department of Cardiology, Odense University Hospital, Odense
  - Department of Cardiology, Viborg Hospital, Viborg

IPD SHARING:
Plan to Share IPD: No